CLINICAL TRIAL: NCT00683514
Title: Oral Vinorelbine And Cisplatin With Concomitant Radiotherapy Followed By Either Consolidation Therapy With Oral Vinorelbine And Cisplatin Plus Best Supportive Care Or Best Supportive Care Alone In Stage III Non Small Cell Lung Cancer (NSCLC), A Randomized Phase III Study
Brief Title: Oral Chemotherapy And Platinum With Radiotherapy Followed Or Not By Consolidation With The Same Chemotherapy In Locally Advanced Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Collaborators: Pierre Fabre Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PM 0259 CA 304 J1
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: NSCLC
Keywords: Untreated locally advanced inoperable stage IIIA or stage IIIB NSCLC amenable to radical radiotherapy to a dose of 66 Gy
MeSH Terms: interventions — Vinorelbine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Other): * cycle 1 & 2 (q 28 days) = chemotherapy : oral vinorelbine (50 mg/m2 d1, d8, d15) and cisplatin (20 mg/m2/d from d1 to d4) combined with radiotherapy
  * cycle 3 & 4 (q 21 days) = chemotherapy : oral vinorelbine (60 mg/m2 d1, d8 for cycle 1, 80 mg/m2 d1 & d8 for cycle 2) and cisplatin (80 mg/m2 d1) plus Best Supportive Care
  Interventions: Drug: Oral Vinorelbine and cisplatin with concomitant radiotherapy 66 Gy (total dose)
- B (Other): * cycle 1 & 2 (q 28 days) = chemotherapy : oral vinorelbine (50 mg/m2 d1, d8, d15) and cisplatin (20 mg/m2/d from d1 to d4) combined with radiotherapy
  * Best Supportive Care only
  Interventions: Drug: Oral Vinorelbine and cisplatin with concomitant radiotherapy 66 Gy (total dose)

INTERVENTIONS:
Drug: Oral Vinorelbine and cisplatin with concomitant radiotherapy 66 Gy (total dose) — q 28 days :
  * 50 mg/m2 oral vinorelbine d1, d8, d15
  * 20 mg/m2/d cisplatin from d1 to d4
Drug: Oral Vinorelbine and cisplatin with concomitant radiotherapy 66 Gy (total dose) — q 21 days :
  * 60 mg/m2 oral vinorelbine d1,d8 for cycle 1 or 80 mg/m2 oral vinorelbine d1,d8 for cycle 2
  * 80 mg/m2 cisplatin d1
  Arms: A

SUMMARY:
This is a multicenter, open-label, randomised, phase III study of 2 cycles of oral vinorelbine in combination with cisplatin concurrently with radiotherapy randomised to either two more cycles of consolidation therapy with oral vinorelbine and cisplatin plus Best Supportive Care (BSC) or BSC alone in patients with unresectable locally advanced non small cell lung cancer (NSCLC).

The primary objective is to compare progression-free survival in both arms, the secondary is to evaluate the response rate, overall survival in both arms, to evaluate the safety profile in both arms and to assess quality of life by the LCSS questionnaire.

ELIGIBILITY:
Main Inclusion Criteria:

* Presence of at least one measurable lesion (RECIST criteria)
* Patients with a Karnofsky Performance Status = or > 80%
* Adequate pulmonary function, bone marrow, hepatic and renal functions

Main Exclusion Criteria:

* Patients with NSCLC stage IV, with NSCLC stages I, II, IIIA (except N2), with NSCLC stage IIIB with tumour extent or pleural effusion
* Symptomatic neuropathy > Grade 1
* Hearing impairment = or > Grade 2
* Concomitant/uncontrolled medical disorder
* Pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2005-04; Primary Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Assessments of measurable and not measurable lesions been carried out at baseline and every 2 treatment cycles by using RECIST criteria | at baseline and every 2 treatment cycles and Regular Follow Up at 2 months intervals during the 1st year after completion of treatment and then every 3 months until progression of the last evaluable patient

SECONDARY OUTCOMES:
Assessment of measurable and not measurable lesions been carried out at baseline and every 2 treatment cycles by using RECIST criteria, LCSS QOL Questionnaire and Physical Examination | At baseline and every 2 treatment cycles, Regular follow up at 2 months intervals during 1 year and then every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Marcello RIGGI, Clinical Development Director, Study Director — Institut de Recherche Pierre Fabre
Locations (1):
- Pierre Fabre Pharma GmbH, Freiburg im Breisgau, Jechtinger Str. 13, Germany